CLINICAL TRIAL: NCT05791760
Title: Effectiveness of Compassion Focused Therapy (CFT) for Reducing Self-criticism in Female Patients with Complex PTSD: a Single-case Experimental Study
Brief Title: The Effectiveness of CFT for Reducing Self-criticism in Patients with Complex PTSD: a Single-case Experimental Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Twente (Other)
Responsible Party: Principal Investigator, Jannis Kraiss, Assistant professor, Principal Investigator, University of Twente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTwente
Record Dates: First submitted 2023-03-13; First posted 2023-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD, Shame, Compassion, Well-being
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Compassion-focused therapy (CFT) (Experimental)
  Interventions: Behavioral: Compassion-focused therapy (CFT) for complex PTSD

INTERVENTIONS:
Behavioral: Compassion-focused therapy (CFT) for complex PTSD — The group protocol includes 12 two-hour sessions. Each session begins and ends with a practical exercise (calming rhythmic breathing) and each session includes psychoeducation (conceptualization, self-compassion). At the end of the session, participants are asked to practice at home between sessions (1 hour per week). The protocol consisted of 3 parts; sessions 1-5 focused on compassion understanding, including psychoeducation on emotion regulation, self-compassion skills, and mindfulness skills. Sessions 6-8 focused on motivation to care, compassion from others, the compassionate self, and the relationship between the compassionate self and self-criticism. Sessions 9-12 focused on using compassion in daily life. The group has a maximum of nine participants and is given by three therapists. All therapists are pre-trained to apply the intervention.

SUMMARY:
PTSD is a mental disorder including psychological symptoms related to severe traumatic event(s). PTSD can negatively affect people's functioning in several life domains. Several effective therapies for the treatment of PTSD have been developed in recent decades. However, these treatments are not effective for every patient. Several studies show that people suffering from PTSD also experience feelings of trauma-related guilt, shame, self-blame and negative self-evaluation. These emotions may contribute to the maintenance cycle of PTSD or even become worse over time. In particularly in patients with trauma who have been exposed to repeated traumatic experiences within the context of interpersonal relationships including childhood sexual/physical abuse and domestic violence. This type of trauma is known as complex PTSD. cPTSD is marked by severe difficulties in problems with self and emotion-regulation, relationship difficulties and shame. One key factor for reducing self-criticism in individuals might be self-compassion as the antidote to self-criticism and shame. Compassion focused therapy by Paul Gilbert focuses specifically on increasing self-compassion. Although some studies show promising results of CFT in patients with cPTSS, the effectiveness for this group has not yet been sufficiently examined. Therefore, this Single case experimental design study is conducted with the primary objective of examining the effectiveness of CFT in reducing the primary outcome self-criticism. Secondary outcomes that will be examined are CFT reduces PTSD symptoms and shame and increases self-compassion and well-being.

This SCED study is a noncurrent multiple baseline across subjects study, consisting of three phases with twice-weekly repeated measurements of self-criticism. First the pre-intervention baseline phase, in which participants are randomly assigned to different baseline lengths (either 5, 6 or 7 weeks). The second phase is the subsequent CFT-intervention, consisting of 12 weeks of weekly CFT group sessions with two-weekly assessments of self-criticism. The third phase is follow up for 5 weeks from the end of the intervention, again including two-weekly assessments of self-criticism. By comparing the baseline phases with the intervention and follow-up phases for individual participants, the effectiveness of the CFT intervention on self-critical beliefs can be determined. Changes that occur within participants can be seen as evidence of intervention effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* The participant is between 18 and 65 years old.
* Diagnosis of cPTSD and severe problems with self criticism (as diagnosed by an experienced clinican).
* The participant gives consent to participate in the study using the online informed consent procedure.
* Sufficient Dutch language proficiency and average intelligence.
* The participant has an e-mail address and is in possession of a smartphone or tablet with access to the internet.
* The participant is willing to complete twice-weekly questionnaires for up to 24 weeks.

Exclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-criticism | Up to 24 weeks
  Measured with the Forms of Self-Criticizing/Attacking and Self-Reassuring Scale (FSCRS-SF). It contains 14 items and is a valid and sensitive measurement scale with adequate psychometric properties including structural validity, convergent validity and sensitivity to change. Higher scores indicate more self-criticism and more self-reassurance. Mean scores range from 0 to 4.

SECONDARY OUTCOMES:
PTSD symptoms | Posttest (T1); 3 months after baseline
  The Post Traumatic Checklist Scale (PCL-5) measures the extent in which participant's experienced PTSD symptoms in the past month. It contains 20 items and is a valid and reliable questionnaire for screening and assessing PTSD in clinical practice. Higher scores indicate more PTSD symptoms. Total scores range from 0 to 80.
Self-compassion | Posttest (T1); 3 months after baseline
  Self compassion will be measured with the Self-Compassion Scale-Short Form (SCS-SF). The SCS-SF contains 12 items. Higher scores reflect higher levels of self-compassion. The Dutch version of the SCS-SF has adequate psychometric qualities. Mean scores range from 0 to 5.
Well-being | Posttest (T1); 3 months after baseline
  The 14-item Mental Health Continuum-Short Form (MHC-SF) measures well-being. Higher scores indicate more well-being. The MHC-SF has shown very good psychometric properties in previous studies. Mean scores range from 0 to 5.
Shame | Posttest (T1); 3 months after baseline
  Experiences of Shame Scale (ESS) is the version of Andrews' Experience of Shame Scale (ESS). The ESS distinguishes between characteristic, behavioral and physical shame. The test consists of 25 statements related to shame. Mean scores rang from 1 to 4 with higher scores indicating more Shame.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No